CLINICAL TRIAL: NCT01419093
Title: A Communication Intervention for Physical Activity in Underserved Communities
Brief Title: Communication Intervention Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5K07CA126985 (NIH); 5K07CA126985 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-17 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Physical Activity
Keywords: Physical Activity; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5A Communication (No Intervention): Behavioral: 5 A intervention for physical activity
  Interventions: Other: 5 A communication intervention

INTERVENTIONS:
Other: 5 A communication intervention — This study will examine the effect of primary care clinicians' communication intervention linked to a community-based exercise program. We will use the 5As in discussion of physical activity in 371 office visits in an ethnically diverse, primarily low income patient population. Secondary and exploratory aims are to provide pilot information on [feasibility and sustainability of the intervention from the patients' and clinicians' perspective and derive effect sizes on the intervention's effect on objective changes in physical activity in a subset of participants.
  Other Names: ethnically diverse physical activity clinician communication

SUMMARY:
The project is a two-arm randomized clinical trial to pilot the feasibility of a communication training intervention for primary care clinicians, linked to a community program referral, on use of the 5As to promote physical activity in underserved patients.

DETAILED DESCRIPTION:
This study will focus on training clinicians to communicate effectively using the 5As and patient-centered communication skills (Aim 1). When implemented fully, the intervention will also include referral to a community fitness program. Clinicians will be randomly assigned to two groups (1 and 2). Group 1 will participate in the training intervention first; group 2 will act as a wait-list control for Group 1. The primary outcome, the effectiveness of the intervention on clinician use of the 5As during routine office visits, will be measured by examining 371 audio-recorded patient visits prior to, immediately, after, and 6 months after the clinician is trained. Secondary outcomes include whether the communication training intervention improved patients' perceived competence to adopt physical activity (Aim 2)and whether clinicians believe that the communication intervention addressed pertinent barriers to promoting exercise (Aim 3). Exploratory outcomes (Aim 4) will [assess potential mediators of the intervention's effect, examine the effect of the intervention on actual physical activity levels in a subset of participants, and create a taxonomy of communication markers for each of the 5As.]

ELIGIBILITY:
Inclusion Criteria:

* Current patients at Westside Health Services
* Be scheduled for a routine, follow-up or health maintenance office visit
* Be practicing clinicians (physicians, physician asst. or nurse practitioner

Exclusion Criteria:

* Have life-threatening acute medical problem which precludes participation
* Unable to read and understand English
* Already achieving recommended level of physical activity
* Planning to move or relocate (clinicians) to another practice in the study period
* Serving as study investigators, consultants, or advisors

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of A's used per visit per discussion of physical activity | 5 years
  The mean 5A Score of patients from clinicians who complete the communicatin interventon will be higher thant the mean 5A Score of patients from physicisns that have not been trained. Analytic plan: Unadjusted analysis will use two-sample t-tests to compare means. Adjusted analyses will use linear mixed effects models as described in the Statistical Analysis section.

SECONDARY OUTCOMES:
Patient-centered Communication Constructs | 5 years
  Patient survey; fifteen items.Assesses patient perceptions of providers' being autonomy supportive versus controlling. Measures participants' feelings of competence at carrying out a treament regimen. Scored by trained coder listening to audiorecorded visits. Clinicians survey; 20 items such as whether the clinician would recmmend the intervention to other clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Carroll, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Westside Health Services, Rochester, New York, United States

REFERENCES:
- [Derived] Carroll JK, Winters PC, Sanders MR, Decker F, Ngo T, Sciamanna CN. Clinician-targeted intervention and patient-reported counseling on physical activity. Prev Chronic Dis. 2014 May 29;11:E89. doi: 10.5888/pcd11.130302. PMID 24874781
- [Derived] Carroll JK, Fiscella K, Epstein RM, Sanders MR, Winters PC, Moorhead SA, van Osch L, Williams GC. Physical activity counseling intervention at a federally qualified health center: improves autonomy-supportiveness, but not patients' perceived competence. Patient Educ Couns. 2013 Sep;92(3):432-6. doi: 10.1016/j.pec.2013.06.031. Epub 2013 Aug 7. PMID 23932756